CLINICAL TRIAL: NCT06087900
Title: Effects of Different Exercise Modalities on Apnea-Hypopnea Index and Oxidative Stress in Patients With Obstructive Sleep Apnea.
Brief Title: Effect of Different Exercise Modalities Training in Patients With Obstructive Sleep Apnea.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EX PHYSIO SPSC 8
Record Dates: First submitted 2023-09-15; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-09

CONDITIONS: Obstructive Sleep Apnea
Keywords: HIIT; Pulmonary function; Sleep; Exercise; Polysomnography
MeSH Terms: conditions — Sleep Apnea, Obstructive; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Moderate continuous training (MICT) (Experimental): The participants received a moderate continuous training (MICT) program of walking or running a treadmill 3 days/week, 12 weeks. This training comprises 5 minutes of warm up at 50-55% of maximal heart rate, following by 50 minutes of exercise at 65-70% of maximal heart rate, and 5 minutes of cool down at 50-55% of maximal heart rate. The intensity of exercise increases to 70-75% of maximal heart rate at week 7-12.
  Interventions: Other: Moderate continuous training (MICT)
- High intensity interval training (HIIT) (Experimental): The participants received a 7x2 high intensity interval training (HIIT) program of walking or running a treadmill 3 days/week, 12 weeks. This training comprises training comprises 5 minutes of warm up at 50-55% of maximal heart rate, following by 28 minutes of exercise (2 minutes of high intensity at 85-90% of maximal heart rate interval with 2 minutes of low intensity at 50-55% of maximal heart rate 7 times), and 5 minutes of cool down at 50-55% of maximal heart rate. The intensity of exercise at high intensity increases to 90-95% of maximal heart rate at week 7-12.
  Interventions: Other: High intensity interval training (HIIT)
- Inspiratory muscle training (IMT) (Experimental): The participants received Powerbreathe ® ClassicLight in this training program. The IMT group demonstrated the training 8 cycles of 30 breath, 5 days/week with progressive load 50% of maximal inspiratory pressure (MIP) at week 1-3, 60% of MIP at week 4-6, 70% of MIP at week 7-9, and 80% of MIP at week 10-12. Every first day of the week participants had to undergoing load adjustment at laboratory
  Interventions: Other: Inspiratory muscle training (IMT)
- Control (Sham Comparator): The CON group did not have any intervention but usual care.
  Interventions: Other: Control

INTERVENTIONS:
Other: Moderate continuous training (MICT) — The participants received a moderate continuous training (MICT) program of walking or running a treadmill 3 days/week, 12 weeks. This training comprises 5 minutes of warm up at 50-55% of maximal heart rate, following by 50 minutes of exercise at 65-70% of maximal heart rate, and 5 minutes of cool down at 50-55% of maximal heart rate. The intensity of exercise increases to 70-75% of maximal heart rate at week 7-12.
  Arms: Moderate continuous training (MICT)
Other: High intensity interval training (HIIT) — The participants received a 7x2 high intensity interval training (HIIT) program of walking or running a treadmill 3 days/week, 12 weeks. This training comprises training comprises 5 minutes of warm up at 50-55% of maximal heart rate, following by 28 minutes of exercise (2 minutes of high intensity at 85-90% of maximal heart rate interval with 2 minutes of low intensity at 50-55% of maximal heart rate 7 times), and 5 minutes of cool down at 50-55% of maximal heart rate. The intensity of exercise at high intensity increases to 90-95% of maximal heart rate at week 7-12.
  Arms: High intensity interval training (HIIT)
Other: Inspiratory muscle training (IMT) — The participants received Powerbreathe ® ClassicLight in this training program. The IMT group demonstrated the training 8 cycles of 30 breath, 5 days/week with progressive load 50% of maximal inspiratory pressure (MIP) at week 1-3, 60% of MIP at week 4-6, 70% of MIP at week 7-9, and 80% of MIP at week 10-12. Every first day of the week participants had to undergoing load adjustment at laboratory
  Arms: Inspiratory muscle training (IMT)
Other: Control — The CON group did not have any intervention but usual care.
  Arms: Control

SUMMARY:
The objective of this study was to compare different exercise modalities (moderate continuous intensity training, high intensity interval training, and inspiratory muscle training) on Apnea-Hypopnea index and oxidative stress in patients with Obstructive sleep apnea.

DETAILED DESCRIPTION:
Forty patients with OSA aged 20 and 50 years old, dividing into 4 groups (MICT, HIIT, IMT, and CON) by stratified (with sex, age, and OSA severity) and single random sampling. The MICT group received 50 minutes of running at 65-70% of maximum heart rate 3 days/week for 12 weeks. The HIIT groups received 28 minutes of running (High intensity at 85-90% of maximum heart rate 2 minutes interval with low intensity 50-55% of maximum heart rate 2 minutes) 3 days/week for 12 weeks. The IMT group received Powerbreathe ® device, performing 240 breath (8 sets) per day at 50% of Maximal inspiratory pressure (MIP), 5 days/week for 12 week. The CON group did not have any intervention but usual care. Data collection was split 2 days (1st day for polysomnography evaluation, and 2nd day for questionnaire, blood collection, body composition, exhaled nitric oxide, pulmonary function, respiratory muscle strength and aerobic capacity). All variables were measured before and after exercise program.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with mild (AHI 5-15) or moderate (AHI 15-30) OSA, aged between 20 - 50 years.
2. BMI between 18.5 - 24.9 kg/ m2.
3. No history of exercise more than 150 min/week for 4 weeks.
4. No used CPAP or discontinue at least 2 weeks.
5. No history for surgery for OSA treatment. Screened by physician that patients have not had Uncontrolled diabetes (blood sugar 180 mg/dL) Uncontrolled hypertension (BP 139/89 mmHg) Any coronary artery disease Any neuromuscular disease Chronic Obstructive Pulmonary Disease; COPD Any cognitive disease Other sleep-related disorders Cancer

7. Not a person with current smoker, menopause or pregnancy. 8. Stable medication. 9. Willing to participate in this research.

Exclusion Criteria:

1. Cannot participate at least 80% of exercise program.
2. Inevitable event (injury, sickness, etc.)
3. Unwilling to continue this research.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Forty patients with OSA aged 20 and 50 years old, dividing into 4 groups (MICT, HIIT, IMT, and CON) by stratified (with sex, age, and OSA severity) and single random sampling.
Enrollment: 40 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-07-09 (Actual)

PRIMARY OUTCOMES:
Apnea-Hypopnea index (event/hr) | Change from Baseline Apnea-Hypopnea index at 12 weeks.
  The study performed polysomnography in the sleep laboratory using standard EEG with frontal leads (F1, F2), central leads (C3, C4), occipital leads (O1, O2), and reference leads at mastoids (M1, M2). Electromyography and electrooculography were also used. Oxygen saturation (SpO2) was measured using a finger probe. Air flow was measured using two methods: a nasal pressure transducer and an oral-nasal thermocouple. Respiratory movements of the thorax and abdomen were monitored using respiratory inductance plethysmography. The position of the body was measured using a position sensor attached to the anterior chest wall on the thoracic belt.
Oxidative stress | Change from Baseline Oxidative stress at 12 weeks.
  Blood was collected into sterile ethylenediaminetetraacetic acid (EDTA) tubes from the cubital vein by a nurse at Exercise Physiology laboratory, Chulalongkorn University. The collected blood was analyzed by a medical technologist. To obtain plasma, the EDTA blood samples were centrifuged at 3,000 rpm for 10 minutes. All plasma samples were stored at a temperature of -80°C until they were used for various assays.
The Pittsburgh Sleep Quality Index (PSQI) | Change from Baseline Sleep-related and Quality of Life by The Pittsburgh Sleep Quality Index (PSQI) questionnaire at 12 weeks.
  The Pittsburgh Sleep Quality Index (PSQI) Thai version was evaluated at baseline and post-intervention to assess subjective sleep quality over the previous 2 weeks. This index aimed to evaluate their subjective sleep quality over the preceding two weeks. The PSQI provided seven component scores, which included assessments of sleep quality, the time taken to fall asleep, the duration of sleep, the regularity of sleep, disturbances during sleep, the use of sleep medications, and daytime dysfunction. By summing up the scores from these subscales, a global score ranging from 0 to 21 was calculated. A global score above 5 is generally considered an indication of poor sleep quality.
The Short Form-36 (SF-36) questionnaire | Change from Baseline Sleep-related and Quality of Life by The The Short Form-36 (SF-36) questionnaire at 12 weeks.
  The Short Form-36 (SF-36) questionnaire Thai version was evaluated at baseline and post-intervention. This questionnaire consists of 36 questions that are used to assess quality of life (QoL) across eight domains related to both physical and mental health. These domains include physical functioning, role limitations due to physical health (role-physical), bodily pain, general health, vitality, social functioning, role limitations due to emotional health (role-emotional), and mental health. Each domain is scored on a scale of 0 to 100, where higher scores indicate a better health-related quality of life (HRQL) compared to lower scores.
The Functional Outcomes of Sleep Questionnaire (FOSQ) | Change from Baseline Sleep-related and Quality of Life by The Functional Outcomes of Sleep Questionnaire (FOSQ) at 12 weeks.
  The Functional Outcomes of Sleep Questionnaire (FOSQ) Thai version was evaluated at baseline and post-intervention. This questionnaire specifically designed to assess health-related quality of life in relation to sleep disorders. It comprises 30 items that examine five domains related to normal daily life: general productivity (8 items), vigilance (7 items), social outcome (2 items), activity level (9 items), and sexual relationship (4 items). Each subscale and a global score were calculated, with the subscale scores ranging from 1 to 4 and the global score ranging from 5 to 20. A lower score indicates a higher level of dysfunction or poorer quality of life.
The Epworth sleepiness scale (ESS) | Change from Baseline Sleep-related and Quality of Life by The Epworth sleepiness scale (ESS) Questionnaire at 12 weeks.
  The Epworth sleepiness scale (ESS) Thai version was evaluated at baseline and post-intervention. This questionnaire is used to assess excessive daytime sleepiness (EDS). The questionnaire consists of eight scenarios where individuals rate their potential for dozing off or falling asleep on a scale of 0 to 3. The ESS has demonstrated excellent internal consistency and test-retest reliability, making it suitable for assessing the effectiveness of interventions. A total ESS score greater than 10 indicates the presence of EDS and a high risk of sleep-related breathing disorders.

SECONDARY OUTCOMES:
Pulmonary function (Forced vital capacity; FVC) | Change from baseline FVC at 12 weeks.
  The participants were instructed to sit on a chair and wear a nose clip. The researcher provided them with a detailed set of instructions to ensure they performed the maneuver correctly according to guidelines of the American Thoracic Society (ATS). Prior to demonstrating forced inspiration and expiration, the participants were asked to perform three cycles of slow normal breathing as part of the FVC maneuver. FVC will be reported in liter (L).
Pulmonary function (Forced Expiratory Volume in one second; FEV1) | Change from baseline FEV1 at 12 weeks.
  The participants were instructed to sit on a chair and wear a nose clip. The researcher provided them with a detailed set of instructions to ensure they performed the maneuver correctly according to guidelines of the American Thoracic Society (ATS). Prior to demonstrating forced inspiration and expiration, the participants were asked to perform three cycles of slow normal breathing as part of the FVC maneuver. FEV1 (L) will be reported in liter (L).
Pulmonary function (The ratio of the forced expiratory volume in the first one second to the forced vital capacity of the lungs; FEV1/FVC) | Change from baseline FEV1/FVC at 12 weeks.
  The participants were instructed to sit on a chair and wear a nose clip. The researcher provided them with a detailed set of instructions to ensure they performed the maneuver correctly according to guidelines of the American Thoracic Society (ATS). Prior to demonstrating forced inspiration and expiration, the participants were asked to perform three cycles of slow normal breathing as part of the FVC maneuver. FEV1/FVC will be reported in percent (%).
Pulmonary function (Peak expiratory flow; PEF) | Change from baseline PEF at 12 weeks.
  The participants were instructed to sit on a chair and wear a nose clip. The researcher provided them with a detailed set of instructions to ensure they performed the maneuver correctly according to guidelines of the American Thoracic Society (ATS). Prior to demonstrating forced inspiration and expiration, the participants were asked to perform three cycles of slow normal breathing as part of the FVC maneuver. PEF will be reported in liter per minute (L/min).
Pulmonary function (Forced expiratory flow at 25 - 75% of FVC; FEF25-75%) | Change from baseline FEF25-75% at 12 weeks.
  The participants were instructed to sit on a chair and wear a nose clip. The researcher provided them with a detailed set of instructions to ensure they performed the maneuver correctly according to guidelines of the American Thoracic Society (ATS). Prior to demonstrating forced inspiration and expiration, the participants were asked to perform three cycles of slow normal breathing as part of the FVC maneuver. FEF25-75% will be reported in liter per second (L/sec).
Pulmonary function (Maximal voluntary ventilation; MVV) | Change from baseline MVV at 12 weeks.
  The participants were instructed to sit on a chair and wear a nose clip. The researcher provided them with a detailed set of instructions to ensure they performed the maneuver correctly according to guidelines of the American Thoracic Society (ATS). During the MVV maneuver, participants were instructed to demonstrate in rapid and forceful inhalation and exhalation for a duration of 10 seconds. MVV will be reported in liter per minute (L/min).
Respiratory muscle strength | Change from baseline Respiratory muscle strength at 12 weeks.
  Respiratory muscle strength was evaluated by measuring Maximal Inspiratory Pressure (MIP) and Maximal Expiratory Pressure (MEP) in centimeters of water (cmH2O). The participants were seated and utilized a portable handheld mouth pressure meter (MicroRPM), along with a nose clip. To assess MIP, participants were instructed to exhale until they emptied their lungs at the point of functional residual capacity (FRC). Participants held the device to their mouth and forcefully inhaled for 1-2 seconds. For the measurement of MEP, participants were directed to inhale until their lungs were completely filled with air, starting from the total lung capacity (TLC) point. Participants were asked to maintain the device on their mouth and forcefully exhaled for 1-2 seconds.
Exhaled nitric oxide (ppb) | Change from baseline Exhaled nitric oxide at 12 weeks.
  The participants were instructed to sit upright and hold the device (NObreath, BedFont, UK). They were asked to take a deep breath and fill their lungs completely, and then exhale through the mouthpiece while ensuring that the ball in the flow indicator remained in the middle of the white band. The exhalation time was set at 12 seconds. Each participant was requested to repeat the measurement three times.
Aerobic capacity (ml/kg/min) | Change from baseline Aerobic capacity at 12 weeks.
  Participants were prepared for a 4-lead electrocardiogram before undergoing exercise tests on a treadmill equipped with a gas analyzer. The protocol began at an intensity of approximately 2 METs and involved increments in speed and/or grade every 20 seconds, equivalent to 0.3 METs. During the last 20 seconds of each 3-minute segment, the speed and grade settings matched those of the standard Bruce protocol (e.g., 3 minutes: 1.7 mph, 10% grade). Heart rate measurements were taken during the last 5 seconds of every minute and at peak exercise. Participants were asked to rate their perceived exertion during the last 5 seconds of each minute and immediately after the test (peak rating of perceived exertion). Blood pressure was measured during the last 30 seconds of minutes 3, 6, 9, and 11, as well as immediately after the test.

CONTACTS AND LOCATIONS:
Overall Officials: Wannaporn Tongtako, Principal Investigator — Chulalongkorn University
Locations (1):
- Faculty of Sports Science, Chulalongkorn University, Pathum Wan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Karlsen T, Nes BM, Tjonna AE, Engstrom M, Stoylen A, Steinshamn S. High-intensity interval training improves obstructive sleep apnoea. BMJ Open Sport Exerc Med. 2017 Feb 8;2(1):bmjsem-2016-000155. doi: 10.1136/bmjsem-2016-000155. eCollection 2016. PMID 29616142
- [Result] Kline CE, Crowley EP, Ewing GB, Burch JB, Blair SN, Durstine JL, Davis JM, Youngstedt SD. The effect of exercise training on obstructive sleep apnea and sleep quality: a randomized controlled trial. Sleep. 2011 Dec 1;34(12):1631-40. doi: 10.5665/sleep.1422. PMID 22131599
- [Result] Nobrega-Junior JCN, Dornelas de Andrade A, de Andrade EAM, Andrade MDA, Ribeiro ASV, Pedrosa RP, Ferreira APL, de Lima AMJ. Inspiratory Muscle Training in the Severity of Obstructive Sleep Apnea, Sleep Quality and Excessive Daytime Sleepiness: A Placebo-Controlled, Randomized Trial. Nat Sci Sleep. 2020 Dec 2;12:1105-1113. doi: 10.2147/NSS.S269360. eCollection 2020. PMID 33293881
- [Result] Andrade FM, Pedrosa RP. The role of physical exercise in obstructive sleep apnea. J Bras Pneumol. 2016 Nov-Dec;42(6):457-464. doi: 10.1590/S1806-37562016000000156. PMID 28117479
- [Result] Krittayaphong R, Bhuripanyo K, Raungratanaamporn O, Chotinaiwatarakul C, Chaowalit N, Punlee K, Kangkagate C, Chaithiraphan S. Reliability of Thai version of SF-36 questionnaire for the evaluation of quality of life in cardiac patients. J Med Assoc Thai. 2000 Nov;83 Suppl 2:S130-6. PMID 11194004